CLINICAL TRIAL: NCT00217022
Title: A Randomized, Double-Blind, Placebo Controlled Trial of Budesonide for the Treatment of Active Lymphocytic Colitis
Brief Title: Budesonide Versus Placebo for the Treatment of Lymphocytic Colitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study closed early, because of low enrollment.
Sponsor: Mayo Clinic (Other)
Collaborators: AstraZeneca (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Darrell S. Pardi, M.D., Physician, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1132-03; IRUSBUEN0002 (Other: AstraZeneca); UL1RR024150 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Lymphocytic Colitis; Diarrhea
Keywords: Lymphocytic Colitis; diarrhea; budesonide
MeSH Terms: conditions — Colitis, Lymphocytic; Diarrhea | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Active Comparator): 9 mg daily
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): three tablets daily
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo, 3 tablets daily
  Arms: Placebo
Drug: Budesonide — 9 mg daily (three tablets)
  Other Names: Entocort EC
  Arms: Budesonide

SUMMARY:
Patients will receive budesonide or placebo for the treatment of active lymphocytic colitis. This study includes stool collections, blood draws, weekly questionnaires and a sigmoidoscopy. The study hypothesis is that budesonide will be safe and effective compared with placebo for the treatment of diarrhea in lymphocytic colitis.

DETAILED DESCRIPTION:
Microscopic colitis is an increasingly diagnosed cause of chronic diarrhea, with two main subtypes: collagenous and lymphocytic colitis. Uncontrolled reports have suggested that various drugs can be beneficial in treating microscopic colitis, but few treatments have been evaluated in randomized controlled trials. Thus, treatment is guided mostly by anecdotal reports, case series, and physicians' experience. In our uncontrolled experience, corticosteroids are one of the most effective therapies for microscopic colitis, but are not typically used as a first line therapy because of toxicity. Budesonide has been reported to be of clinical benefit in small, uncontrolled series of patients with microscopic colitis, and recent controlled trials showed that it is superior to placebo in collagenous colitis. We propose a study of budesonide in patients with the lymphocytic type of microscopic colitis.

Patients will have stool specimen and blood drawn at the start of the study. Patient will take either Budesonide or placebo for 8 weeks. At the end of treatment, patient will have stool collection and sigmoidoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea, defined as greater than 4 bowel movements per day and greater than "mild"; currently on no treatment or active despite treatment.
* Lymphocytic colitis confirmed histologically within one year of enrollment

Exclusion Criteria:

* Previous unsuccessful treatment with corticosteroids or immunosuppressive drugs
* History of severe corticosteroid side effects
* Corticosteroid, ticlopidine, or flutamide use within the previous 4 weeks
* Antibiotic, mesalamine or bismuth subsalicylate use within two weeks
* Current use of anticholinergics, cholestyramine, narcotics, ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, erythromycin, or grapefruit juice
* Known active medical conditions, including cancer, infection, uncontrolled hypertension or diabetes, osteoporosis, peptic ulcer disease, glaucoma, cataracts, liver cirrhosis or history of tuberculosis
* Other diarrheal conditions (sprue, infection, hyperthyroidism, lactose intolerance)
* Pregnant or nursing females
* Patients without a telephone or unable to communicate in English over the telephone, or unable or unwilling to give consent
* Known hypersensitivity to or intolerance of budesonide.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell S. Pardi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mayo Clinic, Rochester, Minnesota from June 2003 - February 2008.
Period: Overall Study
Arm/Group | Budesonide | Placebo
Started | 12 | 4
Completed | 11 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide | Placebo | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (19) | 59 (12) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Satisfactory Control of Diarrhea During at Least Three of the Last Four Weeks
Description: Subjects were asked if they felt they had satisfactory control of their diarrhea, along with the number of stools and type of stool (loose, water, formed, hard) the patient were experiencing. The rating of "satisfactory control" of diarrhea was therefore a partially subjective measure. This outcome measure was to be recorded for three out of the last four weeks that a subject was on the study; subjects were to take part in the study approximately 8 weeks.
Time Frame: Three out of last four weeks that the subject was on the study
Measure: Number; unit: participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 11 | 4
participants | 11 | 4

2. Secondary Outcome: Histologic Improvement in Post Treatment Colon Biopsies Compared to Baseline Biopsies
Description: The histopathology scoring system included epithelial damage, lamina propria cellularity and intraepithelial lymphocytosis, each scored on a four point scale ("normal" (0), "mildly increased" (1), "moderately increased" (2), "severely increased" (3)).
Time Frame: Baseline (day 1 of study) and at eight weeks (approximately)
Population: Only 8 of the subjects on the budesonide arm returned for the biopsy, so only those subjects on that arm were analyzed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Budesonide | Placebo
Number analyzed (Participants) | 8 | 3
participants | 7 | 1

ADVERSE EVENTS:
Arm/Group | Budesonide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 0/11 | 0/4

LIMITATIONS AND CAVEATS:
Study closed early, because of low enrollment. Primary physician for patients with lymphocytic colitis would prescribe Budesonide off label for them. Subjects not interested in placebo trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT00217022/Prot_SAP_ICF_000.pdf